CLINICAL TRIAL: NCT01878058
Title: Identifying Prostate Brachytherapy Seeds Using MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 12-5302-CE
Record Dates: First submitted 2012-10-23; First posted 2013-06-14 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer Patients Who Have Brachytherapy Seed Implant
Keywords: Prostate cancer; Brachytherapy; Seed implant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI Scan (Other): Patients will receive an extra MRI scan in addition to their routine scan.
  Interventions: Other: MRI Scan

INTERVENTIONS:
Other: MRI Scan — Patient will receive an additional MRI scan in addition to their standard of care imaging

SUMMARY:
This study will look at the feasibility of using a type of Magnetic Resonance Imaging called Susceptibility Weighted Imaging (SWI) to detect your implanted radioactive seeds. Researchers hope that using SWI will eliminate the need to use CT imaging to detect your implanted radioactive seeds.

This study will also see if the MRI seed detection is as effective as current standard practice of seed detection (routine MRI and CT imaging). This technique would be beneficial for brachytherapy without the need to fuse the MRI and CT images, as is done currently.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Histologic diagnosis of adenocarcinoma of the prostate
3. No contraindications for Pelvic body MRI
4. Patients undergoing LDR brachytherapy at PMH and scheduled for post implant analysis with CT-MR (standard at PMH)
5. Ability to provide written informed consent to participate in the study

Exclusion Criteria:

1. Contraindication for Pelvic body MRI
2. Patient not willing/consenting for this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Determine if using the MR scan -(SWI) used to detect the implanted radioactive seeds will reduce registration errors | 6 months
Determine if using the MR scan -(SWI) used to detect the implanted radioactive seeds will reduce planning time for the post-implant plan | 6 months
Determine if using the MR scan -(SWI) used to detect the implanted radioactive seeds will eliminate the CT scan of the patient. | 6 months

SECONDARY OUTCOMES:
Compare the differences in MR seed identification using the MR pulse sequence vs. CT images. | 6 months
  Our goal is to perfectly match these two modalities with acceptance test of 97%. This technique would be beneficial for LDR (Low Dose Rate) Brachytherapy without need to fuse the CT and MR images and eliminate any image registration uncertainly.

OTHER OUTCOMES:
Compare the prostate dosimetry (V100 and D90) in prostate low dose rate therapy using MR alone with CT/MR fusion. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Saibishkumar Elantholiparameswaran, MD, Principal Investigator — University Health Network, The Princess Margaret
Locations (1):
- University Health Network, The Princess Margaret, Toronto, Ontario, Canada